CLINICAL TRIAL: NCT06185855
Title: A Simplified Approach to Predicting the Malignancy of Breast Lesions: Nomogram in Ultrasonography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Lixin Jiang, Chief Physician, RenJi Hospital
Other Study IDs: LY2023-210-B
Record Dates: First submitted 2023-12-16; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer Diagnosis; Breast Cancer
Keywords: Breast cancer diagnosis; Mammographic model; Breast disease; Clinical decision-making; Quantitative analysis
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malignant: Malignant Breast Lesion Group: This group would include patients diagnosed with breast cancer who have undergone breast lesion surgery and had preoperative ultrasound examinations at the hospital.
  Interventions: Other: Retrospective Ultrasonographic Data Analysis
- Benign: Benign Breast Lesion Control Group: This group would consist of patients with benign breast lesions, who also underwent breast lesion surgery and had preoperative ultrasound examinations.
  Interventions: Other: Retrospective Ultrasonographic Data Analysis

INTERVENTIONS:
Other: Retrospective Ultrasonographic Data Analysis — The intervention involves a detailed retrospective analysis of ultrasonographic data from patients who underwent breast lesion surgery. The study focuses on developing a quantitative nomogram model, which integrates patient age and significant sonographic characteristics of breast lesions. The purpose is to differentiate breast lesions and assess their malignancy in a non-invasive, accurate manner. This analysis uses data collected from January 2020 to June 2023, including clinical and ultrasound examination records from patients who met the inclusion criteria. The intervention does not involve any direct patient interaction or new diagnostic procedures.

SUMMARY:
This study aims to construct and validate a quantitative mammographic model based on breast ultrasound images, incorporating patient characteristics such as age and significant sonographic features. The model is intended for precise discrimination of breast lesions while assessing its diagnostic performance in clinical practice. Our goal is to provide a reliable adjunct tool to enhance the clinical decision-making of healthcare professionals and potentially improve early screening and accurate diagnosis of breast diseases.

DETAILED DESCRIPTION:
Data Collection: This study retrospectively collected clinical and ultrasound examination data from patients who underwent breast lesion surgery at our hospital from January 2020 to June 2023. Inclusion criteria included patients with complete clinical information and available ultrasound image data. Parameters extracted from this data included age, 2D ultrasound images, Doppler ultrasound images, and ultrasound diagnostic reports. Feature extraction from ultrasound images included 2D lesion information (maximum diameter, orientation, echogenicity, morphology, margins, calcification type, ductal changes), Doppler information (blood flow pattern, resistance index), and BI-RADS classification based on suspicious ultrasound findings by physicians.

Model Development: Firstly, we conducted multicollinearity analysis using Variance Inflation Factor (VIF) to select variables with VIF less than 5, aiming to reduce the impact of collinearity. We used post-operative pathological results of breast lesions as the gold standard for model development. In the R programming language, we utilized the caret package to randomly split the final samples into training and validation sets in a 7:3 ratio based on the outcome variable (benign or malignant breast lesions) while setting a random seed (set.seed) for result reproducibility. Subsequently, we performed univariate logistic regression analysis on binary variables in the training set, retaining variables with P < 0.05, followed by multivariate logistic regression analysis to identify independent predictors of breast lesion malignancy.

Model Validation: To validate the model's performance, we constructed a nomogram based on the weight allocation of each independent predictor. Then, we comprehensively validated the model in the validation set, including calculating sensitivity, specificity, accuracy, and concordance. Receiver Operating Characteristic (ROC) curves were plotted, and the area under the curve (AUC) was calculated to determine the optimal threshold for quantitatively predicting the probability of breast cancer occurrence in patients. Additionally, we performed Decision Curve Analysis (DCA) to assess the net clinical benefit of the model at different patient decision thresholds. DCA helps determine the practical utility of the model in clinical decision-making and identifies the optimal threshold for predicting the probability of disease occurrence, aiding physicians in making better decisions. These validation metrics were used to evaluate the model's performance, accuracy, and potential application in real clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent breast lesion surgery at Renji Hospital affiliated with Shanghai Jiao Tong University School of Medicine during the specified period (January 2020 to June 2023).
* Patients who had a preoperative ultrasound examination of the breast lesion at the same hospital.
* Availability of complete clinical and ultrasonographic data for the patients.
* Histopathological confirmation of breast lesions post-surgery.

Exclusion Criteria:

* Patients who received neoadjuvant therapy (chemotherapy, targeted therapy, immunotherapy, etc.) prior to surgery.
* Patients diagnosed with metastatic breast malignancy.
* Cases with poor quality or incomplete ultrasound images.
* Patients with a Breast Imaging Reporting and Data System (BI-RADS) category 1 diagnosis.
* Incomplete clinical records or missing critical data relevant to the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients who underwent breast lesion surgery at Renji Hospital, affiliated with Shanghai Jiao Tong University School of Medicine, between January 2020 and June 2023. This population is diverse in terms of age and includes individuals diagnosed with various types of breast lesions, ranging from benign to malignant. All participants had undergone preoperative ultrasound examinations, which are critical for the retrospective analysis in this study.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the Ultrasonographic Nomogram in Predicting Breast Lesion Malignancy | Retrospective analysis of data collected from January 2020 to June 2023
  The primary outcome measure is the accuracy of the developed nomogram in differentiating between malignant and benign breast lesions. This will be determined by comparing the nomogram's predictions against the actual histopathological findings from breast lesion surgeries. Accuracy will be quantified in terms of sensitivity, specificity, positive predictive value, negative predictive value, and the area under the receiver operating characteristic curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, Principal Investigator — Shanghai Jiao Tong University School of Medicine Affiliated Renji Hospital

IPD SHARING:
Plan to Share IPD: No